CLINICAL TRIAL: NCT00030771
Title: Preoperative Chemoradiotherapy vs. Chemotherapy Alone in Non-small Cell Lung Cancer (NSCLC) Patients With Mediastinal Lymph Node Metastases (Stage IIIA, N2): A Randomized Prospective Phase III Trial
Brief Title: Preoperative Chemoradiotherapy vs. Chemotherapy Alone in NSCLC Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 16/00; SWS-SAKK-16/00 (Other: SAKK); EU-20138
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
Keywords: squamous cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; adenosquamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Neoadjuvant Chemoradiotherapy + Chemotherapy + Surgery
  Interventions: Drug: Chemotherapy; Radiation: Radiotherapy; Procedure: Surgery
- Arm B (Active Comparator): Neoadjuvant Chemotherapy + Surgery
  Interventions: Drug: Chemotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: Chemotherapy — Docetaxel (Taxotere®) 85 mg/m2 1 hour iv infusion d1 Cisplatin 100 mg/m2 1 hour iv infusion d1 Schedule: 3 cycles repeated every 21 days
Radiation: Radiotherapy — Radiotherapy (3 weeks after last chemotherapy administration) 44 Gy in 22 fractions concomitant boost technique in 3 weeks
  Arms: Arm A
Procedure: Surgery — 3-4 weeks after termination of radiotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and cisplatin, use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving chemotherapy with radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. It is not yet known if chemotherapy plus radiation therapy is more effective than chemotherapy alone before surgery in treating non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying docetaxel and cisplatin with or without radiation therapy to see how well they work when given before surgery in treating patients with stage IIIA non-small cell lung cancer that has spread to lymph nodes in the chest.

DETAILED DESCRIPTION:
The main objective of this trial is to compare feasibility and efficacy of sequential neoadjuvant chemoradiotherapy with 44 Gy concomitant boost to neoadjuvant chemotherapy alone.

Secondary objectives are to assess the value of PET in predicting pathological response and eventfree survival in stage IIIA NSCLC, and a health economic analysis of the two regimens. Further to compare the amount of serum DNA in patients with stage IIIA, pN2 NSCLC before chemotherapy, before surgery and at the second follow-up visit (i.e. four months after surgery or treatment failure for patients who can not be operated) in patients randomized into the trial SAKK 16/00 and to correlate the DNA variation with tumor response, remission duration and overall survival.

OUTLINE: This is a prospective randomized phase III trial. Patients are stratified according to mediastinal bulk (5 cm or more vs less than 5 cm), weight loss in the past 6 months (5% or more vs less than 5%), and participating center. Patients are randomized to 1 of 2 treatment arms.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Squamous, adenosquamous, large cell, or poorly differentiated
* Stage IIIA (T1-3, N2, M0)

  * N2 disease confirmed by 1 of the following:

    * Mediastinoscopy
    * Bronchoscopy with fine-needle aspiration or esophagoscopy

      * All N3 lymph nodes must be negative by positron-emission tomography (PET) AND CT scan (< 1 cm in the largest diameter)
    * PET scan

      * Both the primary tumor and at least 1 N2 lymph node must be positive in PET scan
      * At least 1 of the PET scan positive N2 lymph nodes is positive in the CT scan (> 1 cm in the largest diameter)
      * All N3 lymph nodes negative in PET scan

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* AST/ALT no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* Cardiac function normal
* No unstable cardiac disease requiring treatment
* No congestive heart failure
* No angina pectoris even if medically controlled
* No significant arrhythmia
* No myocardial infarction in the past 3 months

Pulmonary:

* Lung function appropriate

Neurologic:

* No history of significant neurologic or psychiatric disorders
* No psychotic disorders
* No dementia
* No seizures

Other:

* No other prior or concurrent malignancies except nonmelanoma skin cancer, adequately treated carcinoma in situ of the cervix, or any other neoplastic disease with a disease-free interval ≥ 5 years
* No active uncontrolled infection
* No uncontrolled diabetes mellitus
* No gastric ulcers
* No pre-existing peripheral neuropathy greater than grade 1
* No contraindications to corticosteroids
* No other serious underlying medical condition that would preclude study participation
* No socioeconomic or geographic condition that would preclude study participation
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior cytostatic chemotherapy

Endocrine therapy:

* No concurrent prednisone except for treatment of acute hypersensitivity reactions or chronic low-dose treatment initiated more than 6 months prior to study entry (i.e., no greater than 20 mg methylprednisolone or equivalent)

Radiotherapy:

* No prior radiotherapy to chest

Surgery:

* Not specified

Other:

* At least 30 days since participation in another clinical study
* No other concurrent experimental drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2001-04-04 (Actual); Primary Completion 2014-04-09 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 1 month after surgery
  Time from randomization to relapse/progression/second tumor/death, whichever occurs first (for all randomized patients). If no event is observed, the patients will be censored at the last time they were known to be alive.

SECONDARY OUTCOMES:
Postoperative mortality assessed | 1 month after surgery
  All deaths occurring within 30 days of the thoracic surgery to remove the primary tumor
Toxicity (hematological, renal and neurological toxicities, nausea and vomiting, weight changes as well as esophageal toxicities) | During treatment
  Assessed according to the NCIC-CTG Expanded Common Toxicity Criteria grading. Special attention shall be given to hematological, renal and neurological toxicities, nausea and vomiting, weight changes as well as esophageal toxicities.
Complete resection rate after surgery | 1 month after surgery
  Assessed according to the NCIC-CTG Expanded Common Toxicity Criteria grading.
Objective response rate measured after completion of chemoradiotherapy | 43 days
  Response rate will be evaluated according to the
  1. WHO response criteria
  2. TNM classification after surgery.
Operability | 1 month after chemo
  Patients who are able to undergo radical resection of their lung cancer after neoadjuvant therapy, as assessed by the thoracic surgeon.
Overall survival | Life-long follow-up until death of patient (up to 30 years)
  Calculated from randomization to the date of death from any cause. Patients not experiencing an event will be censored at the last time they were known to be alive.
Failure pattern | Life-long follow-up until death of patient (up to 30 years)
  Defined as location of first tumor progression or relapse. Failure can be local relapse (area of primary tumor or mediastinum), distant relapse (all others) or the combination thereof.

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Pless, MD, Study Chair — Kantonsspital Winterthur KSW; Hans-Beat Ris, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois; Diana Naehrig, MD, Principal Investigator — Universitaetsspital-Basel; Roger Stupp, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudoise
Locations (25):
- Germany (2):
  - Klinik Loewenstein gGmbH, Löwenstein
  - Klinikum der Stadt Mannheim, Mannheim
- Serbia (2):
  - Institut za plucne bolesti, Kamenitz
  - Institute of Oncology, Kamenitz
- Switzerland (21):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Kantonsspital, Baden
  - Saint Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Bruderholz, Bruderholz
  - Kantonsspital Graubuenden, Chur
  - Kantonsspital Freiburg, Fribourg
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Pluridisciplinaire d' Oncologie, Lausanne
  - Kantonsspital Liestal, Liestal
  - Kantonsspital Olten, Olten
  - FMH Onkologie/Haematologie, Rheinfelden
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital, Thun
  - Kantonsspital Winterthur, Winterthur
  - Onkozentrum, Zurich
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tieu BH, Sanborn RE, Thomas CR Jr. Neoadjuvant therapy for resectable non-small cell lung cancer with mediastinal lymph node involvement. Thorac Surg Clin. 2008 Nov;18(4):403-15. doi: 10.1016/j.thorsurg.2008.07.004. PMID 19086609
- [Derived] Pless M, Stupp R, Ris HB, Stahel RA, Weder W, Thierstein S, Gerard MA, Xyrafas A, Fruh M, Cathomas R, Zippelius A, Roth A, Bijelovic M, Ochsenbein A, Meier UR, Mamot C, Rauch D, Gautschi O, Betticher DC, Mirimanoff RO, Peters S; SAKK Lung Cancer Project Group. Induction chemoradiation in stage IIIA/N2 non-small-cell lung cancer: a phase 3 randomised trial. Lancet. 2015 Sep 12;386(9998):1049-56. doi: 10.1016/S0140-6736(15)60294-X. Epub 2015 Aug 11. PMID 26275735